CLINICAL TRIAL: NCT05842070
Title: The Stanford Egg Freezing Study: Investigating a Low-Cost, Low-Intensity Oocyte Cryopreservation Protocol
Brief Title: The Stanford Egg Freezing Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Ruth Bunker Lathi, Professor of Obstetrics & Gynecology, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69100
Record Dates: First submitted 2023-04-06; First posted 2023-05-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Fertility Issues; Reproductive Issues
Keywords: Access-to-care; Low-cost; Egg freezing; Fertility preservation; Oocyte cryopreservation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: A non-inferiority margin of -5 MIIs per retrieval was selected based on existing literature on planned OC, which reports expected yields of 9-13 MIIs with approximately 45% variability in ovarian stimulation response (per literature). Setting the margin at -5 ensured that observed differences in oocyte yield would be beyond expected variation, while still maintaining clinical viability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Intensity Protocol (Experimental): Participants choose the low-cost, low-intensity egg-freezing protocol
  Interventions: Procedure: Low-Intensity Egg Freezing Protocol
- High-intensity protocol (Active Comparator): Participants choose a routine high-intensity egg-freezing protocol
  Interventions: Procedure: High-Intensity Egg Freezing Protocol

INTERVENTIONS:
Procedure: Low-Intensity Egg Freezing Protocol — The low-intensity egg freezing protocol involves fewer ultrasounds, bloodwork and injections, contributing to a lower cost. Otherwise, this protocol does not differ significantly from the other routine high-intensity clinic protocols.
  Other Names: Cardinal Protocol
  Arms: Low-Intensity Protocol
Procedure: High-Intensity Egg Freezing Protocol — The high-intensity egg freezing protocol is a routinely used clinic protocol where patients are coming for frequent ultrasounds and bloodwork, as well as more injections, contributing to a higher overall cost for egg-freezing.
  Arms: High-intensity protocol

SUMMARY:
The purpose of this study is to see if the investigators can obtain non-inferior clinical outcomes (similar numbers of oocytes) using the Cardinal protocol, a cost-conscious, low-intensity egg freezing protocol, compared to other routinely used high-intensity clinic protocols. This is a new program for Stanford's Fertility Clinic, so the investigators are assessing patient experience and cost-benefit of a low-cost, low-intensity approach that has demonstrated non-inferiority in IVF for infertility treatment, but has not been similarly evaluated in egg freezing. All enrolled participants will choose the Cardinal protocol or the routine high-intensity protocol designated by their physician. The investigators will then assess number of eggs retrieved, as well as patient satisfaction, cost, and time needed off work to complete the egg freezing cycle. The study's findings could ultimately open the door to implementation of lower-cost standardized protocols that would be more affordable and accessible to people who may otherwise not be able to pursue fertility preservation.

DETAILED DESCRIPTION:
The 2020-2025 strategic plan of ASRM lists equitable, affordable access to reproductive healthcare as a high-focus priority goal, with a pressing need to identify cost-effective treatments that patients shut out by finances can still afford. While there have been some efforts made to broaden access to infertility treatment with in-vitro fertilization (IVF), there are very limited efforts to do for patients desiring egg freezing as a strategy for deferred reproduction. The Stanford Egg Freezing Study is a novel clinical trial that will be assessing for non-inferiority of outcomes from a low-cost, low-intensity approach called the Cardinal Protocol, compared to the routinely used high-intensity clinic protocols. Participant enrollment will occur locally in the greater Bay Area from patients pursuing egg freezing for fertility preservation at Stanford's Fertility clinic.

To specifically review the Cardinal Protocol, this is a low-cost, low-intensity egg-freezing protocol designed to be cost-conscious and streamlined compared to all the other routine protocols used in clinic. This means medication doses are protocolized, decreasing the total number of injections and medications needed, bloodwork and ultrasounds are limited, prevention of premature ovulation is done using oral progestins, and trigger timing is standardized as opposed to timed by provider preference, resulting in a projected cost-savings of on average $5,800 ($3,700-$11,000). This protocol has been reviewed and approved by all 8 REI board-certified infertility specialists at Stanford who based on the literature and practice deem this a standard protocol that could be offered to patients interested in a lower-cost approach.

The investigators hypothesize that the Cardinal protocol compared to the other routinely used high-intensity clinic protocols, will offer non-inferior clinical outcomes for patients with respect to the number of eggs retrieved, improve overall patient satisfaction, and decrease out-of-pocket costs, as well as time required off work to complete the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ovary-bearing individuals of reproductive age 18-40, interested in pursuing OC
* AMH > 0.3 ng/mL
* AMH < 7 ng/mL

Exclusion Criteria:

* AMH > 7 ng/mL or physician concern for risk of developing severe OHSS
* History of severe OHSS
* Severe diminished ovarian reserve (DOR) def. as AMH < 0.3 ng/mL or FSH > 15
* BMI > 45
* Any contraindications to ovarian stimulation or outpatient egg retrieval under anesthesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Mature oocytes cryopreserved per egg freezing cycle | Identified within 24-48 hours of the oocyte retreival
  Number of mature oocytes cryopreserved
Oocyte yield per retrieval or egg freezing cycle | Identified within 24 hours of the oocyte retreival
  Number of oocytes retrieved

SECONDARY OUTCOMES:
Participant satisfaction with egg freezing experience and specific protocol (assessed using the Likert scale) | Identified on post-cycle survey completed 1-2 months following oocyte retrieval
  Assessment of satisfaction on scale of 1-5 towards egg freezing process and protocol
Out-of-pocket costs of the egg freezing cycle for the participant | Identified on post-cycle survey completed 1-2 months following oocyte retrieval and via the electronic medical record
  With or without insurance coverage for egg freezing, with an assessment of total costs or charges of the cycle, including medication costs
Time off-work needed to complete the egg freezing cycle | Identified on post-cycle survey completed 1-2 months following oocyte retrieval
  Not including the egg retrieval procedure day
Additional cost per additional oocytes retrieved | Identified from post-cycle survey completed 1-2 months following oocyte retrieval
  Cost-benefit analyses

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Lathi, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Fertility and Reproductive Health Services, Sunnyvale, California, United States

IPD SHARING:
Plan to Share IPD: No